CLINICAL TRIAL: NCT01336400
Title: Genome-wide Single Cell Haplotyping as a Generic Method for Preimplantation Genetic Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); Universitair Ziekenhuis Brussel (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Professor Joris Vermeesch, Universitaire Ziekenhuizen Leuven
Other Study IDs: IWT-TBM-090878
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Preimplantation Genetic Diagnosis
Keywords: Single cell haplotyping; Preimplantation genetic diagnosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA, single blastomere DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PGD-FISH: Following couples opting for preimplantation genetic diagnosis on the basis of FISH:
  * couples suffering a complex chromosomal rearrangement (CCR)
  * couples with X-linked recessive disorders
  * couples that carry a balanced chromosomal rearrangement
  Interventions: Other: single cell haplotyping
- PGD-PCR: Following couples opting for preimplantation genetic diagnosis on the basis of PCR:
  -couples at risk for the transmission of monogenic diseases
  Interventions: Other: single cell haplotyping

INTERVENTIONS:
Other: single cell haplotyping — We aim to collect single blastomeres from spare IVF embryos of 30 couples to optimize and test methods for single cell haplotyping. We aim to collect 20 and 10 couples coming to the fertility centre for FISH- or PCR-based PGD respectively. In both groups, at least 5 different indications for PGD will be collected. Per couple, we will perform 10 SNP-arrays: 2 for the couple donating the embryo, 4 for family members (often parents of the couple) and 4 for blastomeres since we aim to pick 2 cells from 2 embryos per couple. For five couples, 2 blastomeres of all available embryos will be aspirated to validate and optimize the phasing methods. Finally, for some embryos, all blastomeres will be picked to be able to prove the reproducibility of single cell haplotyping.

SUMMARY:
The investigators previously developed approaches to SNP-, CNV- and haplo-type single human cells (Vanneste et al. 2009, Nature Medicine). These methods open the possibility to be developed into a novel generic diagnostic technique which broadens the spectrum of disease-alleles that can be selected against during preimplantation genetic diagnosis (PGD) and which enables to help those couples that cannot be supported by PGD yet. PGD is the genetic analysis of a single blastomere from an in vitro fertilized (IVF) embryo and it is offered to couples to avoid the transmission of heritable genetic disorders to their offspring. PGD analyses are performed for (1) autosomal dominant or recessive monogenic diseases, (2) X-linked disorders and (3) chromosomal aberrations that may result in aneuploid conceptions. This novel method is likely to outperform and hence, replace current techniques for preimplantation genetic diagnosis. In this project the investigators will bring the technology from a proof-of-principle to the clinical application. To this end the investigators will make computational improvements for accurate single blastomere SNP-, CNV- and haplo-typing and perform a large validation study. For the validation studythe investigators will analyse the genomes of the blastomeres derived from 60 spare embryos of different origin: (1) Embryos diagnosed as genetically abnormal using current PCR- and FISH-protocols. (2) Embryos diagnosed as normal for the investigated region using current PCR- and FISH-protocols, but not of sufficient quality to be transferred or frozen. (3) Embryos of the sex that is selected against following PGD based sex-selection, or embryos of the sex that is selected for but of insufficient quality to be transferred or frozen. (4) Embryos that were not biopsied in a PGD cycle since they suffer a slight growth delay. This validation study will allow us to evaluate (1) the clinical validity (false positive and negative rate) and (2) clinical applicability (in terms of ease of use, success rate, etc.). In addition, it will bring us essential further fundamental insights in the origins and mechanisms of chromosomal instability operating during early embryogenesis and its consequences for clinical applications of PGD. Finally, following the validation study, this project will clinically implement the technique to treat 10 families.

ELIGIBILITY:
Inclusion Criteria:

Blastomeres biopsied from spare embryos ((A) Embryos diagnosed as genetically abnormal using current PCR- and FISH-protocols; (B) Embryos diagnosed as normal for the investigated region using current PCR- and FISH-protocols, but not of sufficient quality to be transferred or frozen; (C) Embryos of the sex that is selected against following PGD based sex-selection, or embryos of the sex that is selected for but of insufficient quality to be transferred or frozen; (D) Embryos that were not biopsied in a PGD cycle since they suffer a slight growth delay.) derived from following patient groups:

1. The first patient group involve couples suffering a complex chromosomal rearrangement (CCR), which is defined as a structural chromosomal rearrangement with at least three breakpoints and an exchange of genetic material between two or more chromosomes.
2. The second patient group involve couples with X-linked recessive disorders.
3. The third patient group consists of couples that carry a balanced chromosomal rearrangement - a translocation, insertion or inversion - that may result in recurrent miscarriage or aneuploid, severely handicapped offspring.
4. A fourth patient group are couples at risk for the transmission of monogenic diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We aim to collect spare embryos of 30 couples that opt for preimplantation genetic diagnosis (see Eligibility Criteria).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joris R Vermeesch, Professor, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Thierry Voet, Professor, Principal Investigator — KU Leuven; Thomas D'Hooghe, Professor, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Yves Moreau, Professor, Principal Investigator — KU Leuven; Karen Sermon, Professor, Principal Investigator — Vrije Universiteit Brussel; De Rycke Martine, Professor, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Vlaams Brabant, Belgium

REFERENCES:
- [Background] Vanneste E, Voet T, Le Caignec C, Ampe M, Konings P, Melotte C, Debrock S, Amyere M, Vikkula M, Schuit F, Fryns JP, Verbeke G, D'Hooghe T, Moreau Y, Vermeesch JR. Chromosome instability is common in human cleavage-stage embryos. Nat Med. 2009 May;15(5):577-83. doi: 10.1038/nm.1924. Epub 2009 Apr 26. PMID 19396175
- [Background] Vanneste E, Voet T, Melotte C, Debrock S, Sermon K, Staessen C, Liebaers I, Fryns JP, D'Hooghe T, Vermeesch JR. What next for preimplantation genetic screening? High mitotic chromosome instability rate provides the biological basis for the low success rate. Hum Reprod. 2009 Nov;24(11):2679-82. doi: 10.1093/humrep/dep266. Epub 2009 Jul 24. PMID 19633308